CLINICAL TRIAL: NCT04436549
Title: Clinical and Pathological Correlations in Chronic Venous Disease
Brief Title: Pathology, Venous Disease, and Clinical Correlations
Acronym: PAVEDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2018.11
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Varicose Veins; Pathology; Symptoms and Signs
Keywords: pathology; varicose veins; chronic venous disease; symptoms
MeSH Terms: conditions — Varicose Veins; Signs and Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with varicose veins: Patients with varicose veins and eligible to receive open surgery (stab avulsion of varicose veins) as routinely care.
  Interventions: Procedure: Stab Avulsion of varicose veins; Diagnostic Test: Histopathologic evaluation of varicose veins

INTERVENTIONS:
Procedure: Stab Avulsion of varicose veins — Stab avulsion is a technique to remove varicose veins. In this procedure, several tiny cuts (incisions) are made in the skin through which the varicosed vein is removed. Removed varicose veins will be collected and analyzed.
  Other Names: Phlebectomy
Diagnostic Test: Histopathologic evaluation of varicose veins — Sample obtained from varicose veins of lower limbs of patients will be collected and immediately fixed in formalin. The tissue fragments will be taken from varicose veins. Subsequently the tissue will be embedded in paraffin and 3-to-4 mm thick sections will be prepared by a microtome. The tissue sections will be processed for histological and immunohistochemical studies of VEGF, MM9, PGP 9.5 AND FRIBRONECTIN. For antibodies the EnVision staining system (Dako EnVision™) will be used. For the analysis of the positive structures detected by immunohistochemistry, a semiquantitative evaluation method will be used.

SUMMARY:
Chronic Venous Disease (CVD) has a high prevalence in the general population of the western world. Varicose veins are the main signs of this disease that are characterized by important pathological vessel wall changes. There are also several symptoms that affect the quality of life of affected patients. The aim of this study is to correlate the main histopathological abnormalities with the type and the intensity of the symptoms.

DETAILED DESCRIPTION:
Chronic Venous Disease (CVD) of the lower limbs is a widespread chronic condition of the western world. There are several signs and symptoms that affect quality of life of patients with CVD. One of the main signs of this disease are varicose veins that are enlarged, swollen, and twisting superficial veins. Vessel wall of varicose veins shows a significant histopathological phenotype, characterized by a distortion of structural architecture: endothelial damage, disorganization of muscle bundles and alteration of the composition of the extracellular matrix (ECM). Symptoms may be different, according to disease state, progression and local inflammatory processes. To date, there is no study that correlate the type and the intensity of symptoms with histopathological phenotype.

Aim of this study is to correlate histopathological phenotype with clinical manifestations.

A cohort of patients with varicose veins scheduled for open surgical treatment that will undergo to stab avulsion of varicose veins will be recruited. Subsequently, venous tissue from stab avulsion will collected in order to evaluate the following biomarkers: VEGF (Vascular -Endothelial Growth Factor), PGP 9.5 (Protein Gene Product 9.5), Fibronectin and Matrix Metalloproteinase- 9 (MMP-9).

VEGF has a key role as a regulator of angiogenesis; its expression is highly regulated by hypoxia, in this case induced by venous hypertension. In addition to being a marker of neoangiogenesis, it increases vascular permeability in inflammatory disorders. PGP 9.5 is a marker of the innervation of the vessel wall that plays an important role in the regulation of venous tone. Fibronectin and MMP-9 are direct markers of ECM remodeling and impairment and they have also a role in chronic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with varicose veins scheduled for surgery

Exclusion Criteria:

* Peripheral artery disease
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with varicose veins that are scheduled to undergo surgery for varicose veins removal.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Expression of Matrix Metalloproteinase-9 (MMP-9) | at 10 month
  EnVision staining system (Dako EnVision™) will be used. A synthetic peptide from the middle region of human MMP9 will be used with dilutions 1:50 with Ethylenediaminetetraacetic acid (EDTA).
Expression of Vascular Endothelial Growth Factor (VEGF) | at 10 month
  EnVision staining system (Dako EnVision™) will be used. Monoclonal mouse Anti-Human vascular endothelial growth factor, code No. M7273 will be used with dilution 1:50 with Ethylenediaminetetraacetic acid (EDTA).
Expression of Fibronectin | at 10 month
  EnVision staining system (Dako EnVision™) will be used. A synthetic peptide made toward the C-terminal region of the human Fibronectin protein (within residues 2250-2300) will be used with dilution 1:400 citrate buffer.
Expression of Protein Gene Product 9.5 (PGP 9.5) | at 10 month
  EnVision staining system (Dako EnVision™) will be used. Purified PGP 9.5 isolated from bovine brain will be used with dilution 1:200 citrate buffer

SECONDARY OUTCOMES:
Correlation of the biomarkers expression with signs and symptoms | At 11 month.
  The expression of the biomarkers that will be studied on venous tissue samples will be correlated with the type of signs and symptoms complained by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., Ph.D., Principal Investigator — University Magna Graecia of Catanzaro
Locations (2):
- Italy (2):
  - CIFL- Interuniversity Center of Phlebolymphology, Catanzaro
  - University Magna Graecia of Catanzaro, Catanzaro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birdina J, Pilmane M, Ligers A. The Morphofunctional Changes in the Wall of Varicose Veins. Ann Vasc Surg. 2017 Jul;42:274-284. doi: 10.1016/j.avsg.2016.10.064. Epub 2017 Mar 11. PMID 28300675
- [Background] Kucukguven A, Khalil RA. Matrix metalloproteinases as potential targets in the venous dilation associated with varicose veins. Curr Drug Targets. 2013 Mar;14(3):287-324. PMID 23316963
- [Background] Kolano P, Bednarski IA, Lesiak A, Skibinska M, Stasikowska-Kanicka O, Danilewicz M, Narbutt J. Overexpression of cathepsin K and vascular endothelial growth factor in chronic venous ulcerations. Postepy Dermatol Alergol. 2020 Apr;37(2):234-239. doi: 10.5114/ada.2020.94840. Epub 2020 May 6. PMID 32489360